CLINICAL TRIAL: NCT00120757
Title: Efficacy of Alendronate Versus Placebo in the Treatment of HIV-1 Associated Osteoporosis, a Multicenter, Randomized, Controlled Trial. ANRS 120 Fosivir
Brief Title: Efficacy of Alendronate Versus Placebo in the Treatment of HIV-associated Osteoporosis (ANRS120)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-002002-30; ANRS120 Fosivir
Record Dates: First submitted 2005-07-11; First posted 2005-07-19 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Osteoporosis; HIV Infections
Keywords: Osteoporosis
MeSH Terms: conditions — Osteoporosis; HIV Infections | interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Alendronate

SUMMARY:
Osteopenia and osteoporosis are being described more frequently in people with HIV infection. This study will test the efficacy of alendronate in comparison with a placebo after 2 years, in people with primary osteoporosis. People will receive the recommended adequate intake of calcium and vitamin D.

DETAILED DESCRIPTION:
The purposes of this trial are:

* To study the efficacy of alendronate in HIV-associated osteoporosis
* To measure the prevalence of osteoporosis in HIV patients and to detect risk factors in a large cohort of HIV patients from the screening phase

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant
* Non menopausal women
* Total femur BMD below -2.5 SD (T score) or lumbar spine BMD below -2.5 SD (T score) or BMD below -1 associated with a vertebral osteoporotic fracture (diminution of vertebral height over 20%)
* HIV infection known for at least 5 years
* CD4 cell count over 50/mm3
* Karnofsky score over or equal to 70
* Written informed consent.

Exclusion Criteria:

* Osteoporosis resulting from a cause other than HIV: vitamin D deficiency (in that case, after receiving high-dose calcium and vitamin D for 1 month, patients will be randomized without a new screening), renal failure, heart failure (NHYA class III or IV), treatment with glucocorticoid at a dose over or equal to 0.5mg/kg/d for 15 days or more at time of inclusion or during the previous 6 months; thyroid or other endocrine disease if untreated for more than 6 months; hypercalciuria
* Testosterone below normal if treatment is hormonal
* BMI below or equal to 18
* Severe lung failure
* Chronic alcohol intoxication
* Ongoing opportunistic infection
* Gastric ulcer of disease interfering with oesophageal motility in the previous 3 months
* History of treatment for osteoporosis
* History of malignancy in the previous 5 years (except skin cancer and Kaposi)
* Cytotoxic chemotherapy or cytokine therapy
* Liver cirrhosis
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2004-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Percentage of variation of lumbar BMD on DEXA scan at month 24 versus month 0 for patients included with lumbar osteoporosis (femoral for those included with only femoral osteoporosis)

SECONDARY OUTCOMES:
Percentage of variation of femoral T-score between M0 and M24
Percentages of variation of lumbar and femoral T score between M0 and M12
Evolution of bone metabolism markers
Occurrence of fractures
Tolerance of alendronate
Measure of the prevalence of osteopenia and osteoporosis in HIV-infected men and women
Description of the evolution of osteoporosis in HIV-infected men and women receiving calcium and vitamin D to define risk factors for osteoporosis in HIV-infected persons

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Rozenberg, MD, Principal Investigator — Hopital Pitie-Salpetriere Paris service de Rhumatologie; Dominique Costagliola, Study Chair — Inserm U720
Locations (3):
- France (3):
  - Service de Medecine Interne hopital Avicenne, Bobigny
  - Service de Rhumatologie hopital Pitie-Salpetriere, Paris
  - Hôpital Necker service des Maladies Infectieuses, Paris

REFERENCES:
- [Derived] Rozenberg S, Lanoy E, Bentata M, Viard JP, Valantin MA, Missy P, Darasteanu I, Roux C, Kolta S, Costagliola D; ANRS 120 Fosivir Study Group. Effect of alendronate on HIV-associated osteoporosis: a randomized, double-blind, placebo-controlled, 96-week trial (ANRS 120). AIDS Res Hum Retroviruses. 2012 Sep;28(9):972-80. doi: 10.1089/AID.2011.0224. Epub 2012 Mar 23. PMID 22353022